CLINICAL TRIAL: NCT04273685
Title: Cognitive Remediation and Social Recovery in Early Psychosis
Acronym: CReSt-R
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Gary Donohoe, Professor, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUIreland3
Record Dates: First submitted 2020-01-30; First posted 2020-02-18 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Psychosis
Keywords: Early Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a feasibility study with a randomised, controlled, outcome-assessor-blind, parallel- group design.
Who Masked: Outcomes Assessor
Masking Description: A randomisation procedure for group allocation will be compiled with an independent statistician. A research assistant, blinded to allocation, will complete outcome assessments at the three time points (Prior to the study commencing, 2 weeks post study completion and follow up at 3 months).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition (Experimental): Cognitive remediation training, cognitive behavioural therapy, social recovery therapy
  Interventions: Behavioral: Cognitive remediation training, social recovery therapy
- Control Condition (Active Comparator): Treatment as usual (TAU),non-directive counselling
  Interventions: Other: treatment as usual

INTERVENTIONS:
Behavioral: Cognitive remediation training, social recovery therapy — 10 weeks cognitive remediation training plus social recovery therapy. One hour face to face contact time with intervention therapist per week. At-home cognitive remediation training completion.
  Arms: Intervention Condition
Other: treatment as usual — 10 weeks Treatment as usual non directive counselling One hour face to face contact time with intervention therapist per week.
  Arms: Control Condition

SUMMARY:
This intervention trial explores the feasibility, effectiveness and acceptability of a novel psycho-social intervention for early psychosis based on a combined cognitive remediation training and cognitive behavioural therapy approach focused on social recovery. The impact of the CReSt-R intervention on social cognition as a primary outcome will be explored in addition to secondary outcome measures such as social and occupational functioning ( Detailed further in this registration). Feasibility of the trial design and the acceptability of the CReSt-R intervention to the target group, 16-35 year olds who are within the first 5 years of a diagnosed psychotic illness, are also explored in this trial.

DETAILED DESCRIPTION:
This study is being carried out as part of a collaborative doctoral award program entitled Youth Mental Health Research Leadership (YOULEAD, www.nuigalway.ie/youlead) and is funded by the Health Research Board, Ireland.

It is a multi centre, randomised pilot study based at the National University of Ireland,Galway with ethical approval from the Galway University Hospital ethical committee. The principal investigator is Prof. Gary Donohoe and study lead Ms. Emma Frawley, both based at the School of Psychology, National University of Ireland, Galway.

Across psychosis spectrum disorders, social cognition is strongly linked to functional outcomes and therefore considered an important target for intervention.Social Cognition is reported to mediate the effects of neurocognition on functional outcomes.This suggests better functional outcomes may be achieved if both neurocognition and social cognition are targeted in intervention and that neurocognitive training alone does not result in significant social cognitive improvements.

People living with experience of psychotic illness often experience barriers to socialising. For example, experience of positive symptoms in schizophrenia can result in psychological challenges and reduced opportunities to meet and engage with other individuals in a social context. In a 2012 review of social cognitive interventions it was concluded that in order to impact higher-order social cognitive processes, there needs to be ample opportunity for practice of skills both in a clinical setting as well as in the community. A recent meta- analysis and meta-regression study also concluded early intervention in psychosis, where there is a multi-component treatment approach, is associated with better outcomes across a number of variables including global functioning and involvement in school or work. Exploration of the feasibility of the CReSt-R intervention and its ability to integrate into a multi-component treatment approach, is integral to this research study.

The CReSt-R study is novel in its approach, combining the CIRCuiTS cognitive training programme, informed by a metacognitive model, with Social Recovery Therapy, informed by cognitive behavioural theory and assertive outreach.

Effectiveness of the intervention will be explored with social cognition and social and occupational function as co primary outcomes. Secondary outcomes of general cognition and social and occupational functioning (Detailed further in this registration). Feasibility of the intervention will be assessed using key indicators of rate of enrollment, blinding effectiveness, rate of retention of participants and completion rate of the primary outcome measures. Acceptability of the intervention will be assessed using the Intrinsic Motivation inventory (IMI) administered on completion of the study and a qualitative study.

When a participant is recruited and consented to the study (via the services they attend) they will be randomised to either an intervention or control group.

In the intervention group the participant will receive 1 hour a week of the CReSt-R intervention for 10 weeks. This will include:

1. Cognitive remediation training (CR). Cognitive remediation training "Is a behavioural training-based intervention that aims to improve cognitive processes [attention, memory, executive function, social cognition, or metacognition] with the goal of durability and generalisability". The programme used in this study is the Computerised Interactive Remediation of Cognition- Training for Schizophrenia (CIRCuiTS). CIRCuiTS is a web based CR programme which targets metacognition, specifically strategy use, in addition to massed practice of cognitive functions (Attention, memory and executive functioning). Collaborative goal setting related to real-world tasks are integral to the programme with the programme tasks and exercises increasing in difficulty in response to the participant's performance and progress. This will be the primary focus of 1:1 therapy for the first 4 weeks with remote practice sessions occurring between therapy visits. After 4 weeks' remote practice will continue and the focus of in-person therapy sessions will bridge to Social Recovery Therapy (SRT) as detailed below.
2. Social Recovery Therapy (SRT) focuses on addressing barriers to individuals interacting in their social environment e.g. social anxiety. It is informed by cognitive behavioural theory and addresses individual goals. It occurs in three stages as defined by the SRT protocol - Stage one focuses on engagement with the participant and collaborative formulation with the purpose of identifying a problem list and establishing a therapeutic relationship. Stage two prepares the participant for new activities with identification of pathways to activity and collaboration with community stakeholders. Stage three promotes engagement in new activities using behavioural experiments to promote social activity. This is the primary focus of in-person therapy sessions from week 5 to 10 alongside remote practice of the CR programme.

In the control group of the study participants will receive Treatment as Usual (TAU) plus 10 weeks of 1:1 non-directive counselling matching the intervention group for time.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 16 and 35 years' old
* History of psychosis: within the first five years of a diagnosed psychotic illness (based on time since first contact with mental health services for a psychotic episode)
* Community-based and clinically stable (in opinion of primary treating team)
* Ability to give consent

Exclusion Criteria:

* History of organic impairment
* History of head injury with loss of consciousness >5-minute duration
* Drug abuse in the preceding 1 month

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Social and Occupational Functional Assessment Scale (SOFAS) (change from baseline) | Post study at 12 weeks and follow up 3-5 months post study
  The Social and Occupational Functional Assessment Scale is a global rating of current functioning ranging from 0 to 100.Lower scores represent lower functioning and higher scores represent higher functioning.For example a score of 100 represents superior functioning in a wide range of activities,a score of 50 represents serious impairment in social, occupational or school functioning, a score of 30 represents an inability to function in almost all areas of activity. The minimum value is 0 and the maximum value is 100.

SECONDARY OUTCOMES:
Time Use Survey | Baseline, post study at 12 weeks,follow up 3-5 months post study
  The Time Use Survey is a semi-structured interview that enquires about time spent over the past month on work, education, voluntary work, leisure, sports, housework or chores, and child care. Time spent on each of the activities is calculated in terms of the average number of hours per week. The activities are summed to create two scores: constructive economic activity (work, education, voluntary work, housework or chores, and child care) and structured activity (constructive economic activity plus leisure and sports activities).A higher score indicates superior social functioning, a lower score represents impaired social functioning. Less than 45 hours of structured activity per week is considered a threshold for being at risk of social disability, less than 30 hours per week is threshold for social disability and indicative of poor social functioning, and less than 15 hours per week is considered to reflect serious social disability.
Cambridge Neuropsychological Test Automated Battery (CANTAB)- Emotion Recognition Task- change being assessed. | Baseline, post study at 12 weeks and 3-5 months post study
  This task measures the ability to identify six basic emotions in facial expressions along a continuum of expression magnitude. Computer-morphed images derived from the facial features of real individuals, each showing a specific emotion, are displayed on the screen, one at a time. Each face is displayed for 200ms and then immediately covered up to prevent residual processing of the image. The participant must select which emotion the face displayed from 6 options (sadness, happiness, fear, anger, disgust or surprise). The task takes 6 minutes to complete.
The Reading the mind in the eyes task- change being assessed. | Baseline, post study at 12 weeks,follow up 3-5 months post study
  This task measures the capacity to understand mental states of others from expressions in the eye region of the face. Participants view 36 photos and choose the most accurate descriptor word from four choices for the thought/feeling that was portrayed. As noted above, definitions of the response choices are embedded in the task. The dependent measure was the total number of correct responses, ranging from 0 to 36
The Hinting Task - change being assessed. | Baseline, post study at 12 weeks,follow up 3-5 months post study
  This task examines the ability to infer the true intent of indirect speech. Ten short passages presenting an interaction between two characters are read aloud. Each passage ends with one of the characters dropping a hint, and participants explain what the character truly meant. If the first response provided was inaccurate, a second hint is delivered, allowing participants to earn partial credit. Total scores range from 0 to 20
The Bell Lysaker Emotion Recognition Task (BLERT)- change being assessed. | Baseline, post study at 12 weeks,follow up 3-5 months post study
  This task measures recognition of seven emotional states: happiness, sadness, fear, disgust, surprise, anger, or no emotion. Participants identified the emotion shown in 21 videos of a male actor providing dynamic facial, vocal-tonal, and upper-body movement cues. Performance Is indexed as the total number of correctly identified emotions (ranging from 0 to 21).
Wechsler abbreviated scale of intelligence- similarities and matrix reasoning subtests | Baseline, post study at 12 weeks,follow up 3-5 months post study
  The similarities and matrix reasoning subtests from the Wechsler Adult Scale of Intelligence 3rd edition (WAIS-III) is a brief, reliable measure of cognitive ability for use in clinical, educational and research settings. The similarities subtests scores range from 0 - 33 with higher scores indicating better verbal comprehension. Matrix reasoning subtest scores range from 0 - 26 with higher scores reflecting better perceptual organization. Once raw scores are derived they are converted to scaled scores adjusted for age.
Wechsler Memory scale 3rd edition- logical memory and letter number sequencing subtests | Baseline, post study at 12 weeks,follow up 3-5 months post study
  The Wechsler Memory Scale 3rd edition, logical memory subtest is used to assess episodic and auditory memory in immediate and delayed conditions.Logical memory immediate scores range from 0-75, and delayed scores range from 0-50.
  The letter-number sequencing subtest from the Wechsler Memory Scale 3rd edition is used to assess working memory. Scores range from 0-21.
  Higher scores on the Wechsler Memory Scale 3rd edition subtests indicate better memory function. Raw scores are converted to scaled scores adjusted for age.
Rey Osterreith Complex Figure (ROCF) | Baseline, post study at 12 weeks,follow up 3-5 months post study
  The Rey Osterreith Complex Figure is an assessment which measures visual memory by asking the participant to reproduce a complicated line drawing, first by copying it freehand and then drawing from memory (immediate and delayed conditions). Scores range from 0-36 with higher scores indicating better visual memory.
STROOP | Baseline, post study at 12 weeks,follow up 3-5 months post study
  The Stroop test measures a person's sustained attention for word reading and color naming with/without interference. A computerized Stroop task measures mean reaction times (RTs) for congruent and incongruent trials. Four colour words (green, red, yellow, and blue) written in congruent or incongruent colour are randomly presented on screen. The Stroop test detects attentional interference via the measurement of response latency (calculated as mean RT for incongruent trials minus mean RT for congruent trials) when participants are asked to inhibit word meaning and indicate the ink colour of the word. Longer latencies are interpreted as greater interference by word content and lower executive function.
The Positive and Negative Symptom Scale (PANSS) | Baseline, post study at 12 weeks,follow up 3-5 months post study
  The Positive and Negative Syndrome Scale (PANSS) is a 30 item scale used to assess symptom severity which includes positive, negative, and general symptom subscales and total scores. Scores range from 7 to 49 for positive and negative symptoms, 16 to 112 for general symptoms, and 30 to 210 for total score. Higher scores indicate higher symptom severity.

OTHER OUTCOMES:
The Intrinsic Motivation Inventory (IMI) | post study at 12 weeks,follow up 3-5 months post study
  The Intrinsic Motivation Inventory is a multidimensional self-report measure of intrinsic motivation intended to assess participant's subjective experience related to a target activity. The instrument can be modified to fit different activities (i.e. therapy). The instrument assesses participant's interest/enjoyment, effort, pressure/ tension, perceived choice and value/usefulness, thus yielding five subscale scores. In the subscales each item is a statement and the participant must indicate the extent to which they agree or disagree with the statement. Item scores range from 1-7 with 1 indicating disagreement and 7 indicating agreement. Subscale scores are calculated by averaging the items scores for the number of items on each subscale. Higher scores indicate more of the concept described in the subscale name.
The Need for Cognition Scale (NCS) | Baseline, post study at 12 weeks,follow up 3-5 months post study
  The Need for Cognition Scale is an 18-item scale that assesses the degree to which participants seek out cognitively challenging activities of daily living and will provide supplementary information to the social and occupational functioning outcome measures. Each item of the scale contains statements relating to cognitive activities and participants must indicate whether or not the statement is characteristic of them or what they do. Item scores range from 1-5 with 1 indicating a statement is extremely uncharacteristic and 5 indicating a statement is extremely characteristic. Item scores are summed with a lowest possible score of -72 and highest score of 72. Higher scores indicate greater tendency to seek out cognitively challenging activities.
Computerised Theory of Mind Task (c-TOM) | Baseline, post study at 12 weeks,follow up 3-5 months post study
  The Computerised Theory of Mind Task is a novel task measuring theory of mind, it is divided into two separate tests: 1. C-TOM Gaze - this test examines eye gaze discrimination using videos of actors making eye movements. 2. C-TOM stories- this test presents short videos of simple stories featuring two characters. This task takes approx. 8 minutes to complete. Scores are measured in terms of number of correct responses (ranging from 0 to 80) with higher scores indicating superior theory of mind ability.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Donohoe, Principal Investigator — National University of Ireland, Galway
Locations (1):
- National University of Ireland, Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bora E, Yucel M, Pantelis C. Theory of mind impairment in schizophrenia: meta-analysis. Schizophr Res. 2009 Apr;109(1-3):1-9. doi: 10.1016/j.schres.2008.12.020. Epub 2009 Feb 4. PMID 19195844
- [Background] Horan WP, Kern RS, Shokat-Fadai K, Sergi MJ, Wynn JK, Green MF. Social cognitive skills training in schizophrenia: an initial efficacy study of stabilized outpatients. Schizophr Res. 2009 Jan;107(1):47-54. doi: 10.1016/j.schres.2008.09.006. Epub 2008 Oct 18. PMID 18930378
- [Background] Kurtz MM, Richardson CL. Social cognitive training for schizophrenia: a meta-analytic investigation of controlled research. Schizophr Bull. 2012 Sep;38(5):1092-104. doi: 10.1093/schbul/sbr036. Epub 2011 Apr 27. PMID 21525166
- [Background] Pinkham AE, Penn DL, Green MF, Buck B, Healey K, Harvey PD. The social cognition psychometric evaluation study: results of the expert survey and RAND panel. Schizophr Bull. 2014 Jul;40(4):813-23. doi: 10.1093/schbul/sbt081. Epub 2013 May 31. PMID 23728248
- [Background] Addington J, Saeedi H, Addington D. Facial affect recognition: a mediator between cognitive and social functioning in psychosis? Schizophr Res. 2006 Jul;85(1-3):142-50. doi: 10.1016/j.schres.2006.03.028. Epub 2006 May 5. PMID 16678388
- [Background] Fett AK, Viechtbauer W, Dominguez MD, Penn DL, van Os J, Krabbendam L. The relationship between neurocognition and social cognition with functional outcomes in schizophrenia: a meta-analysis. Neurosci Biobehav Rev. 2011 Jan;35(3):573-88. doi: 10.1016/j.neubiorev.2010.07.001. Epub 2010 Jul 8. PMID 20620163
- [Background] Joseph J, Kremen WS, Franz CE, Glatt SJ, van de Leemput J, Chandler SD, Tsuang MT, Twamley EW. Predictors of current functioning and functional decline in schizophrenia. Schizophr Res. 2017 Oct;188:158-164. doi: 10.1016/j.schres.2017.01.038. Epub 2017 Jan 28. PMID 28139356
- [Background] Sheridan AJ, Drennan J, Coughlan B, O'Keeffe D, Frazer K, Kemple M, Alexander D, Howlin F, Fahy A, Kow V, O'Callaghan E. Improving social functioning and reducing social isolation and loneliness among people with enduring mental illness: Report of a randomised controlled trial of supported socialisation. Int J Soc Psychiatry. 2015 May;61(3):241-50. doi: 10.1177/0020764014540150. Epub 2014 Jul 7. PMID 25001267
- [Background] Fiszdon JM, Reddy LF. Review of social cognitive treatments for psychosis. Clin Psychol Rev. 2012 Dec;32(8):724-40. doi: 10.1016/j.cpr.2012.09.003. Epub 2012 Sep 21. PMID 23059624
- [Background] Reeder C, Pile V, Crawford P, Cella M, Rose D, Wykes T, Watson A, Huddy V, Callard F. The Feasibility and Acceptability to Service Users of CIRCuiTS, a Computerized Cognitive Remediation Therapy Programme for Schizophrenia. Behav Cogn Psychother. 2016 May;44(3):288-305. doi: 10.1017/S1352465815000168. Epub 2015 May 25. PMID 26004421
- [Background] Fowler D, Hodgekins J, French P. Social Recovery Therapy in improving activity and social outcomes in early psychosis: Current evidence and longer term outcomes. Schizophr Res. 2019 Jan;203:99-104. doi: 10.1016/j.schres.2017.10.006. Epub 2017 Oct 22. PMID 29070442
- [Background] Reeder C, Huddy V, Cella M, Taylor R, Greenwood K, Landau S, Wykes T. A new generation computerised metacognitive cognitive remediation programme for schizophrenia (CIRCuiTS): a randomised controlled trial. Psychol Med. 2017 Nov;47(15):2720-2730. doi: 10.1017/S0033291717001234. Epub 2017 Sep 4. PMID 28866988
- [Background] Green MF, Horan WP, Lee J. Nonsocial and social cognition in schizophrenia: current evidence and future directions. World Psychiatry. 2019 Jun;18(2):146-161. doi: 10.1002/wps.20624. PMID 31059632
- [Background] Green, M. F., & Horan, W. P. (2010). Social Cognition in Schizophrenia. Current Directions in Psychological Science, 19(4), 243-248. https://doi.org/10.1177/0963721410377600
- [Background] Reeder C, Wykes T (2010). Cognitive Interaction Remediation of Cognition - a Training for Schizophrenia (CIRCuiTS). King's College London: UK.
- [Background] Correll CU, Galling B, Pawar A, Krivko A, Bonetto C, Ruggeri M, Craig TJ, Nordentoft M, Srihari VH, Guloksuz S, Hui CLM, Chen EYH, Valencia M, Juarez F, Robinson DG, Schooler NR, Brunette MF, Mueser KT, Rosenheck RA, Marcy P, Addington J, Estroff SE, Robinson J, Penn D, Severe JB, Kane JM. Comparison of Early Intervention Services vs Treatment as Usual for Early-Phase Psychosis: A Systematic Review, Meta-analysis, and Meta-regression. JAMA Psychiatry. 2018 Jun 1;75(6):555-565. doi: 10.1001/jamapsychiatry.2018.0623. PMID 29800949
- [Background] CREW (2012). Deﬁnition of Cognitive Remediation. Cognitive Remediation Expert Working Group: Florence, Italy.
- [Derived] Frawley E, Cowman M, Cella M, Cohen D, Ryan E, Hallahan B, Bowie C, McDonald C, Fowler D, Wykes T, Donohoe G. Cognitive Remediation and Social Recovery in Early Psychosis (CReSt-R): protocol for a pilot randomised controlled study. Pilot Feasibility Stud. 2022 May 24;8(1):109. doi: 10.1186/s40814-022-01064-6. PMID 35610711